CLINICAL TRIAL: NCT05435560
Title: Characterizing the Neuropharmacology of Dexmedetomidine Through Trimodal Imaging
Brief Title: Neurochemical Mechanisms of the Awake vs. Anesthetized Brain
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Boston University (Other)
Responsible Party: Principal Investigator, Christin Y. Sander, PhD, Dr Christin Sander, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2021P003426
Record Dates: First submitted 2022-04-22; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Anesthesia; Healthy
Keywords: Dopamine; Anesthesia; Positron Emission Tomography; Magnetic Resonance Imaging; Electroencephalograpy; Sleep
MeSH Terms: interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (Experimental): During the imaging scan subjects will receive an initial 1µg/kg bolus of dexmedetomidine up to a maximum dose of 80 µg, infused through IV over 10 minutes. After the bolus has been administered, a constant infusion of up to 0.6 µg/kg/hr (0.01 µg/kg/min) of dexmedetomidine will be maintained for the remainder of the scan (about 60 minutes).
  Interventions: Drug: Dexmedetomidine
- Saline (Placebo Comparator): A saline infusion will be used as a placebo comparator for the dexmedetomidine infusion. It will be administered in the same manner and dosages as the dexmedetomidine.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexmedetomidine — During the imaging scan subjects will receive an initial bolus of dexmedetomidine over 10 minutes. After the bolus has been administered, a constant infusion of dexmedetomidine will be maintained for the remainder of the scan (about 60 minutes).
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Saline — During the imaging scan subjects will receive an initial bolus of saline over 10 minutes. After the bolus has been administered, a constant infusion of saline will be maintained for the remainder of the scan (about 60 minutes).
  Arms: Saline

SUMMARY:
The investigators will be studying the sedative drug dexmedetomidine using hybrid PET/fMRI/EEG imaging to better understand the neuropharmacology of anesthesia/artificially induced sleep.

DETAILED DESCRIPTION:
A group of healthy volunteers will undergo simultaneous PET/fMRI/EEG imaging under two different conditions: while being administered a sedative (dexmedetomidine), and while being administered a normal saline infusion, as a control. The order of these two scans will be randomized, and the study design is open label (ie subjects and investigators know which session will be the control scan and which one will be the sedative scan). Investigators hope that by comparing the results of the sedative and control scans, the different neuromodulatory states involved in the transition from wakefulness to medically induced vs naturally occurring sleep can be better understood.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-45.
* No contraindications to MRI or PET scanning.

Exclusion Criteria:

* Contraindications to fMRI scanning and PET scanning (including presence of a cardiac pacemaker or pacemaker wires, metallic particles in the body, vascular clips in the head or previous neurosurgery, prosthetic heart valves, claustrophobia);
* Pregnancy or breast feeding;
* Current or past history of major medical, neurological, or psychiatric condition;
* History of major head trauma;
* Any cardiovascular disorders, including heart disorders or high blood pressure [>155/95];
* Breathing problems such as severe asthma;
* Bleeding disorder, or use of anticoagulants;
* Bladder obstruction, urinary problems, or history of impaired elimination;
* Known kidney or liver problems;
* Intestinal blockage;
* Raynaud syndrome
* Peripheral nerve injury;
* Diabetes;
* Glaucoma;
* Sleep disorder, such as sleep apnea, insomnia, or narcolepsy
* Current use of any drugs that affect sleep
* Current or recent use of medications (neurological or psychiatric) affecting brain function
* Current or past history of chronic pain (assessed at discretion of PI);
* History of allergic reactions
* History of chronic obstructive pulmonary diseases
* Ulcerative skin conditions or other dermatologic conditions which could interfere with blood pressure cuff placement
* Body mass index above 30
* Current smoker
* Lack of current health insurance coverage
* Employed under the direct supervision of the investigators conducting the research
* Hair in dreadlocks, twists, or braids that cannot be removed
* Eczema on the scalp or face

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-12 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Brain positron emission tomography (PET) imaging signals. | 2 hours
  Changes in dopamine receptor availability will be quantified from brain PET images.
Functional magnetic resonance imaging (fMRI) signals. | 2 hours
  fMRI measures of hemodynamic responses.
Differences in electroencephalography (EEG) measures between arousal and anesthesia. | 2 hours
  Arousal states will be characterized from changes in the EEG power spectrum.

SECONDARY OUTCOMES:
Heart rate | 2 hours
  Heart rate variability.
Pulse oximetry | 2 hours
  Amplitude of pulse oximetry signal.
Respiratory physiology | 2 hours
  Breathing rate (breaths per minute).

CONTACTS AND LOCATIONS:
Overall Officials: Christin Y Sander, PhD, Principal Investigator — Athinoula A. Martinos Center for Biomedical Imaging
Locations (1):
- Athinoula A. Martinos Center for Biomedical Imaging, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No